CLINICAL TRIAL: NCT05072977
Title: Prospective Randomised Controlled Study in 2 Parallel Arms Comparing Corneal Haze, Visual and Refractive Outcomes and Postoperative Pain According to the Mode of De-epithelialisation (Laser Versus Manual Alcohol) During Photorefractive Keratectomy
Brief Title: Photorefractive Keratectomy (PRK) : Comparison of Corneal Haze Between Two Modes of De-epithelialisation (Laser Versus Manual Alcohol)
Acronym: H-TransPKR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulty
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASD_2021_8
Record Dates: First submitted 2021-09-29; First posted 2021-10-11 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Myopia; Astigmatism
Keywords: Myopia; Astigmatism; Corneal haze; Trans Photorefractive Keratectomy; Alcohol Photorefractive Keratectomy
MeSH Terms: conditions — Myopia; Astigmatism; Corneal Opacity | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TransPRK (Experimental)
  Interventions: Procedure: TransPRK
- Alcohol PRK (Active Comparator)
  Interventions: Procedure: Alcohol PRK

INTERVENTIONS:
Procedure: TransPRK — A Merocel sponge is soaked in a saline solution to expand before being gently applied to the corneal surface in three gestures similar to painting. This standardised procedure avoids inhomogeneous wetting of the cornea, which would result in uneven ablation. The laser ablation is then performed.
  Arms: TransPRK
Procedure: Alcohol PRK — A ring is placed in the centre of the cornea and filled with 20% alcohol. After 20 seconds of exposure, the alcohol is absorbed with a small sponge and the corneal epithelium is debrided with a polyvinyl alcohol expanding sponge (Merocel, Medtronic). The entire cornea is rinsed with balanced salt solution and the epithelium is peeled away from the corneal stroma. The corneal bed is then dried with a small sponge and laser ablation is performed.
  Arms: Alcohol PRK

SUMMARY:
surgical correction of ametropia. A number of improvements have been introduced to overcome the side effects and complications such as corneal haze, epithelial irregularities induced by wound healing, pain and delayed visual acuity recovery associated with PRK surgery. During traditional PRK, the corneal epithelium is mechanically debrided before stromal ablation is performed. Alcohol PRK is frequently used as an alternative to mechanical epithelial debridement and is considered simpler and faster. Transepithelial PRK (TransPRK) is a new method in which the corneal epithelium is photoablated by the laser in one step using a specific ablation profile.

This study attempts to establish a means of quantitatively and objectively measuring corneal haze, using patented software based on optical coherence tomography (OCT) of the cornea. This will confirm or refute the hypothesis of a lower occurrence of corneal haze after TransPRK (experimental group) versus PRK with alcohol (control group). Each patient will have one eye randomised to one of the two groups being compared.

ELIGIBILITY:
Inclusion Criteria:

* Planned Photorefractive Keratectomy in both eyes
* Simple myopia or myopic astigmatism, refractive spherical equivalent between -0.50 and -9.0 diopters in both eyes with regular corneal topography

Exclusion Criteria:

* Only one eye operated on
* At least one contraindication to refractive surgery, namely : keratoconus, minimum corneal thickness < 400 µm, severe dry syndrome, progressive corneal infection
* Personal history of corneal surgery
* Personal history of ocular pathology other than simple myopia or myopic astigmatism
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Corneal haze assessed with the the software analysing the corneal OCT images | 1 month after refractive surgery
  Corneal haze assessed by the intensity of the luminosity of the whole cornea (expressed as a percentage) evaluated by the software analysing the corneal OCT images.

CONTACTS AND LOCATIONS:
Overall Officials: Alain SAAD, MD, Principal Investigator — Hôpital Fondation A. de Rothschild
Locations (1):
- Hôpital Fondation A. de Rothschuld, Paris, France